CLINICAL TRIAL: NCT05200390
Title: Closing the Gap in Health Disparities and Improving Health Outcomes: Evaluation of a Single Center Expansion of Continuous Glucose Monitor Access in Patients With Type 2 Diabetes
Brief Title: Evaluation of a Single Center Expansion of Continuous Glucose Monitor Access in Patients With Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chieh Chen (Other)
Collaborators: St. John Fisher College (Unknown)
Responsible Party: Sponsor-Investigator, Chieh Chen, Pharmacy Resident - PGY2, State University of New York - Upstate Medical University
Organization: State University of New York - Upstate Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1788320
Record Dates: First submitted 2022-01-06; First posted 2022-01-20 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Type 2 Diabetes
Keywords: continuous glucose monitor; FreeStyle Libre 2; health disparity; pharmacists
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Continuous Glucose Monitor (Experimental): Adult patients with Type 2 Diabetes on any anti-diabetic regimen utilizing continuous glucose monitors for 3 months
  Interventions: Device: Continuous glucose monitor

INTERVENTIONS:
Device: Continuous glucose monitor — FreeStyle Libre 2 system

SUMMARY:
The purpose of this pilot study is to hopefully generate interest that will lead to more robust trials evaluating FreeStyle Libre 2 sensors in patients with type 2 diabetes on any diabetes regimen. Hopefully the trial will ultimately pave the way to future trials that will prompt clinicians, policymakers, and insurers to re-evaluate the current criteria defining the coverage of continuous glucose monitors (CGM).

The objectives of the study are to 1) Determine if there is difference in diabetes control in adult participants with type 2 diabetes before and after management with FreeStyle Libre 2, 2) Compare participant satisfaction with glucose monitoring and diabetes distress in adult participants with type 2 diabetes before and after management with FreeStyle Libre 2 and 3) Compare the frequency of hypoglycemia in adult participants with type 2 diabetes before and after management with FreeStyle Libre 2.

DETAILED DESCRIPTION:
This will be a prospective, single-center, pre-post pilot study where enrolled participants will be given free FreeStyle Libre 2 sensors for 3 months and will be followed by pharmacists in the Upstate Adult Medicine Clinic.

During the first visit, pharmacists will order a baseline hemoglobin A1c, confirm the participant's current medication list, provide CGM education and assess patient's willingness to scan. Participants will also be asked to participate in a voluntary initial satisfaction survey (Glucose Monitoring Satisfaction Survey). Sensors will be placed at the end of the first visit. No medication changes will be made in order to obtain baseline data for each participant. All initial visits will be conducted in-office. Baseline characteristics will be collected at this visit.

The second visit will be scheduled approximately 2 weeks after the initial visit and will also be in-office. Since no medication changes were made during the first visit, the second visit will provide baseline CGM data, which will be reviewed with the participant. All subsequent follow-up visits will be scheduled at 2-week intervals unless an earlier visit is determined to be necessary by the pharmacist. At the discretion of the pharmacists, subsequent follow-up visits can either be a telemedicine encounter or an in-office visit. CGM data and medication changes will be documented at each visit.

The final visit will be scheduled approximately 3 months after sensor placement and will be in-office. Participants will be asked to participate in the post satisfaction survey (Glucose Monitoring Satisfaction Survey). Pharmacists will repeat the hemoglobin A1c, review the final medication list, remove the sensors, and review plan for self-monitoring blood glucose with patient moving forward.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 2 Diabetes with

  1. Hemoglobin A1c above goal 6.5%-8% based on participant specific factors defined in the ADA guidelines (e.g. comorbidities and age) OR
  2. Identified glycemic excursions, including hypoglycemia based on documented blood glucose readings of < 70 mg/dL via point-of-care glucose testing, lab testing or self-monitoring or reported signs and symptoms of hypoglycemia documented in the medical record
* Referred and actively followed by pharmacy for at least 3 months prior to study enrollment
* Have at least one encounter with pharmacist within the last 3 months
* Have at least one A1c documented while under pharmacist care
* On at least one anti-diabetic medication
* Demonstrates willingness (at the discretion of the investigators) to scan the CGM several times a day
* Demonstrates willingness (at the discretion of the investigators) to attend regular office visits or phone calls

Exclusion Criteria:

* Currently pregnant or actively trying to conceive
* Receiving dialysis
* Currently followed by the endocrinology clinic for diabetes
* Current or past CGM use in the last 6 months prior to study enrollment
* Participant meets criteria for insurance coverage of CGM
* Known allergy to medical adhesive
* Wearing any implanted medical device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-01-24 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Change in percent time in range of 70-180mg/dL (%TIR) | From baseline and at 3 months
  Percentage

SECONDARY OUTCOMES:
Change in Glucose Monitoring Satisfaction Survey (GMSS) scores | From baseline and at 3 month
  Numeric number
Change in %TIR | From baseline and at 1 month
  Percentage
Change in %TIR | From baseline and at 2 months
  Percentage
Change in hemoglobin A1c | From baseline and at 3 months
  Percentage
Change in Percent Time Active | From baseline and at 1 month
  Percentage
Change in Percent Time Active | From baseline and at 2 months
  Percentage
Change in Percent Time Active | From baseline and at 3 months
  Percentage
Change in Percent Time Below Range less than 54mg/dL (%TBR <54mg/dL) | From baseline and at 1 month
  Percentage
Change in %TBR <54mg/dL | From baseline and at 2 months
  Percentage
Change in %TBR <54mg/dL | From baseline and at 3 months
  Percentage
Change in Percent Time Below Range less than 70mg/dL (%TBR <70mg/dL) | From baseline and at 1 month
  Percentage
Change in %TBR <70mg/dL | From baseline and at 2 months
  Percentage
Change in %TBR <70mg/dL | From baseline and at 3 months
  Percentage
Change in Percent Time Above Range more than 180mg/dL (%TAR >180mg/dL) | From baseline and at 1 month
  Percentage
Change in %TAR >180mg/dL | From baseline and at 2 months
  Percentage
Change in %TAR >180mg/dL | From baseline and at 3 months
  Percentage
Change in Percent Time Above Range more than 250mg/dL (%TAR >250mg/dL) | From baseline and at 1 month
  Percentage
Change in %TAR >250mg/dL | From baseline and at 2 months
  Percentage
Change in %TAR >250mg/dL | From baseline and at 3 months
  Percentage
Change in Percent Coefficient of Variation (%CV) | From baseline and at 1 month
  Percentage
Change in %CV | From baseline and at 2 months
  Percentage
Change in %CV | From baseline and at 3 months
  Percentage
Percentage of patients at goal %TIR | 1 month
  Percentage
Percentage of patients at goal %TIR | 2 months
  Percentage
Percentage of patients at goal %TIR | 3 months
  Percentage
Percentage of patients at goal % Time Active | 1 month
  Percentage
Percentage of patients at goal % Time Active | 2 months
  Percentage
Percentage of patients at goal % Time Active | 3 months
  Percentage
Percentage of patients at goal %TBR <54mg/dL | 1 month
  Percentage
Percentage of patients at goal %TBR <54mg/dL | 2 months
  Percentage
Percentage of patients at goal %TBR <54mg/dL | 1, 2, and
  Percentage
Percentage of patients at goal %TBR <70mg/dL | 1 month
  Percentage
Percentage of patients at goal %TBR <70mg/dL | 2 months
  Percentage
Percentage of patients at goal %TBR <70mg/dL | 3 months
  Percentage
Percentage of patients at goal %TAR >180mg/dL | 1 month
  Percentage
Percentage of patients at goal %TAR >180mg/dL | 2 months
  Percentage
Percentage of patients at goal %TAR >180mg/dL | 3 months
  Percentage
Percentage of patients at goal %TAR >250mg/dL | 1 month
  Percentage
Percentage of patients at goal %TAR >250mg/dL | 2 months
  Percentage
Percentage of patients at goal %TAR >250mg/dL | 3 months
  Percentage
Percentage of patients at goal % CV | 1 month
  Percentage
Percentage of patients at goal % CV | 2 months
  Percentage
Percentage of patients at goal % CV | 3 months
  Percentage

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Phillips, PharmD, CACP, Principal Investigator — St. John Fisher College
Locations (1):
- Upstate Health Care Center, Syracuse, New York, United States